CLINICAL TRIAL: NCT04679376
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate the Safety and Efficacy of Statins in Adult Patients With Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Statins for the Treatment of NASH
Acronym: STAT NASH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manal F. Abdelmalek, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-007824
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Atorvastatin Treatment (Experimental): Subjects who have a histology-proved NASH with fibrosis stage 2 or higher will receive atorvastatin for 96 weeks
  Interventions: Drug: Atorvastatin
- Group 2: Placebo (Placebo Comparator): Subjects who have a histology-proved NASH with fibrosis stage 2 or higher will receive a placebo for 96 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 40 mg daily administered orally in tablet or capsule form
  Other Names: Lipitor
  Arms: Group 1: Atorvastatin Treatment
Drug: Placebo — Administered daily orally in tablet or capsule form, contains no active medicine
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this research study is to determine whether the study drug, atorvastatin (Lipitor®), is safe and effective in improving the features of NASH.

ELIGIBILITY:
Inclusion Criteria:

* Definite NASH on a liver biopsy obtained ≤ 90 days prior to randomization with a NAFLD activity score (NAS) of ≥ 4 with at least 1 in each component of the NAS according to NASH CRN grading52
* Fibrosis stage ≥ 2 as assessed by liver biopsy
* Not currently on statin therapy
* Provision of written informed consent
* Agree to use of effective contraceptive measures if female of child bearing potential.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from study enrollment: Any chronic liver disease other than NASH (i.e., drug-induced, viral hepatitis, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, hemochromatosis, A1AT deficiency, Wilsons disease)
* Cirrhosis, as assessed clinically or histologically
* Presence of vascular liver disease
* BMI ≤ 25 kg/m2
* Excessive alcohol use (> 20 g/day) within the past 2 years
* AST or ALT > 250 U/L.
* Type 1 diabetes mellitus
* Bariatric surgery in the past 5 years.
* Weight gain of > 5% in past 6 months or > 10% change in past 12 months.
* Inadequate venous access
* HIV antibody positive, hepatitis B surface antigen positive (HBsAg), or HCV RNA positive.
* Receiving an elemental diet or parenteral nutrition
* Chronic pancreatitis or pancreatic insufficiency
* Any history of complications of cirrhosis (i.e. ascites, hepatic encephalopathy, or portal hypertensive bleeding), even if absent or optimized with medical management at time of screening
* Concurrent conditions: a) Inflammatory bowel disease, b) Unstable angina, myocardial infarction, transient ischemic events, or stroke within 24 weeks of screening, c) Ongoing infectious, immune mediated disease within previously 1 years, d) Any malignant disease (other than basal cell carcinoma of the skin) within previous 5 years, e) Prior solid organ transplant, f) Any other concurrent condition which, in the opinion of the investigator, could impact adversely on the subject participating or the interpretation of the study data.
* Concurrent medications including: a) Anti-NASH therapy(s) initiated after the liver biopsy diagnosing NASH. Anti-NASH therapies include S-adenosyl methionine (SAMe), milk thistle, and vitamin E at dose of ≥ 400 IU/day; b) Antidiabetic mediation which may impact NASH histology started in the past 12 months including thiazolidinediones (glitazones), dipeptidyl peptidase 4 inhibitors (gliptins) or glucagon-like peptide 1 analogs; c) Immune modulatory agents including systemic steroids, methotrexate, anti-TNF-α therapies (infliximab, adalimumab, etanercept) or anti-integrin therapy (namixilab).
* Self-reported or known marijuana or illicit drug use 30 days before the screening
* The following laboratory abnormalities within 90 days of screening: a) HbA1C > 9.0%, b) Neutrophil count < 1.0 x 109/L, c) Platelets < 100 109/L, d) Hemoglobin < 10 g/dl, e) Albumin < 3.5 g, f) Prolonged international normalized ratio (INR), g) Any elevation of bilirubin above normal (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction), h) Serum creatinine > 1.5 mg/dl, i) Creatinine clearance ≤ 50 ml/minute calculated by Crockroft-Gault or creatinine > 1.5x upper limit of normal
* Pregnancy or breastfeeding.
* Women, of childbearing age, who are not willing to practice effective contraception (i.e., barrier, oral contraceptives, or past medical history of hysterectomy) for the 48-week duration of the trial and for 1 month after the first administration of the drug.
* Participation in an investigational drug study within past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in NASH as measured by improvement in NAS score Improvement in NAS score (≥ 2 points) with no worsening in fibrosis stage (≥1 point) OR improvement in fibrosis with no worsening of NASH (change in the NAS score of ≤ 0 points). | Baseline, 96 weeks
  One overall score of NASH improvement will be derived from improvement in NAS score OR no worsening in fibrosis.

SECONDARY OUTCOMES:
NASH resolution as measured by (diagnosis by pathologist) (from definite- to not- NASH)..... | Baseline, 96 weeks
  Histological change from NASH to No NASH
Change in fibrosis stage as measured by change in stage | Baseline, 96 weeks
  Ordinal variable
Change in each component of NASH histologic features as measured by presence or ab presence or absence of features or their severity. | Baseline, 96 weeks
  Existing features may improve in severity or disappear as an indication of improvement of NASH.
Change in serum aminotransferase (ALT) and aspartate aminotransferase (AST) levels as measured by plasma concentrations | Baseline, 96 weeks
Change in makers of hepatic fibrosis markers as measured by (FIB-4,51 liver stiffness by Fibroscan®) | Baseline, 96 weeks
Change in capture attention parameter (CAP) score (with Fibroscan®) | Baseline, 96 weeks
Serum creatine phosphokinase (CPK) as measured by serum concentration | Baseline, 96 weeks
Change in serum lipids as measured by serum concentration | Baseline, 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manal Abdelmalek, MD, MPH, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT04679376/ICF_000.pdf